CLINICAL TRIAL: NCT02615015
Title: Single Nucleotide Polymorphisms in the Deoxyribonuclease 1 Gene Impair Its Activity and Are Increased in a ST-elevation Acute Coronary Syndrome Patient Cohort Compared to Healthy Controls
Brief Title: SNPs in the DNase 1 Gene Impair Its Activity and Are Increased in a STE-ACS Patient Cohort Compared to Healthy Controls
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Andreas Mangold, MD, Medical University of Vienna
Other Study IDs: 1947/2014
Record Dates: First submitted 2015-11-12; First posted 2015-11-25 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: Deoxyribonuclease
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood draw, DNA isolation, plasma isolation
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ST elevation myocardial infarction patient cohort: Patients who suffered from ST elevation myocardial infarction since 2006, referred to the General Hospital of Vienna and received primary percutaneous coronary intervention.
  Interventions: Other: Blood draw
- Healthy proband cohort: Age matched healthy individuals who voluntarily participate in the study.
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw

SUMMARY:
Neutrophil extracellular traps (NETs) and deoxyribonuclease (DNase) activity determine outcome in ST elevation acute coronary syndrome (STE-ACS). DNase single nucleotide polymorphisms (SNPs) were increased in a japanese cohort.

In the present study, the investigators seek to measure DNase SNPs frequency in a caucasian STE-ACS cohort compared to healthy controls (each n=400). The investigators will compute polymorphisms, DNase activity, NET surrogate markers and clinical variables in regression models.

DETAILED DESCRIPTION:
Background Acute coronary syndrome (ACS) is among the leading causes of death(1). Atherosclerosis and coronary thrombotic occlusion are driven by inflammatory pathomechanisms(2). The investigators have shown neutrophilic activation and neutrophil extracellular traps (NETs) at the culprit lesion site of ST-elevation ACS (STE-ACS) patients(3). NETs are well described components of thrombi, building a condensation nucleus for platelets, erythrocytes and fibrinogen. NET-containing thrombi can be effectively lysed by deoxyribonuclease (DNase) in vitro(4). By adding DNase, the investigators showed potent acceleration of tissue plasminogen activator-mediated lysis of coronary thrombi ex vivo. Surrogate markers of NETs are strong predictors of acute coronary events(5). In STE-ACS patients, NETs directly correlated with cardiac magnet resonance-measured infarct size. Moreover, increased coronary DNase activity correlated with smaller infarct size(3).

Two major endogenous plasmatic DNases have been described, namely DNase 1 and DNase gamma(6). Several polymorphisms of the gene encoding for DNase 1 affecting its activity are known(7,8). The single nucleotide polymorphism (SNP) Q222R in the DNase 1 gene, leading to impaired extracellular DNase activity, was correlated with increased incidence of myocardial infarction in Japanese patients(9). SNPs associated with reduced DNAse activity are also known for DNase gamma, but no associations with ACS have been investigated. Present data implicate a critical balance between formation and degradation of NETs and outcome of ACS.

Rationale The investigators hypothesize that coronary endoluminal NET formation is a major component of acute macro- and microvessel atherothrombosis. Extracellular DNase degrades NETs, thus down-regulating overwhelming NET formation. Impaired DNase activity increases the risk for ACS. Thus, the investigators seek to test the presence of polymorphisms in the DNase gene impairing DNase activity in a STE-ACS population.

Aims

1. To compare single nucleotide polymorphisms in the DNase 1 and gamma gene in STE-ACS patients, coronary artery disease patients and healthy controls using polymerase chain reaction
2. To test DNase activity in plasma of these patients and healthy controls and to correlate that with the respective gene expression type
3. To test NET formation and NET surrogate markers and to correlate those with DNase activity and DNase SNPs
4. To correlate these data with surrogate markers of infarct size, reperfusion, long term outcome parameters and risk factors for coronary artery disease.

Methods

Patients

The investigators will contact patients (n=400) who have been hospitalized in the General Hospital of Vienna in the past 10 years for ST-elevation acute coronary syndrome undergoing primary percutaneous coronary intervention (pPCI) with TIMI 0-1. These patients will be invited for a consultation. The investigators will perform the following investigations with patients willing to join the study:

* Medical history
* Detailed clinical examination
* Electrocardiography
* Echocardiography
* Routine blood draw
* Blood draw for research experiments Any patient with relevant clinical findings will be led to further diagnostic evaluation. MACE occurring between the acute coronary event until presence will be surveyed at the consultation. All patients will be contacted once a year to assess MACE.

Healthy donors Blood samples from healthy donors (n=400) will be obtained by a peripheral blood draw from the cubital vein. The probands will be recruited by bulletins in the General Hospital of Vienna.

Real time polymerase chain reaction Cells will be lysed and DNAwill be isolated using a DNAeasy kit (Applied Biosystems). DNA or will be analyzed for DNase SNPs using primer/probe assays (Applied Biosystems). The ABI PRISM 7000 Sequence Detection System and software (Applied Biosystems) will be used.

NET surrogate marker determination

Nucleosomes For the detection of DNA-histone complexes (nucleosomes), an ELISA-Cell death detection kit (Roche Diagnostics GmbH, Germany) will be employed. Optical density (OD) values will be normalized to the internal positive control and expressed as arbitrary nucleosome units/ml (NU/ml). The intra-assay positive control equals 1000 NU/ml.

MPO-DNA complexes Myeloperoxidase (MPO)-associated DNA fragments will be identified using a capture ELISA. 96-well microplates will be coated with an anti-MPO monoclonal capturing antibody (ABD Serotec, UK). As detection antibody, the investigators will use a peroxidase labeled anti-DNA monoclonal antibody (Cell Death Detection ELISA Plus Kit, Roche Diagnostics GmbH, Germany). All measurements will be performed in duplicates and values will be specified as mean ODs.

Double stranded DNA For the detection of double stranded DNA (dsDNA) in patient plasma, the investigators will employ a Quant-iT PicoGreen dsDNA Assay (Invitrogen, USA) on 96-well microplates. PicoGreen is a fluorescent nucleic acid stain for the quantification of dsDNA in solution. Fluorescence will be measured by a Varioskan Flash microplate reader (Thermo Scientific, USA) and normalized to the provided standard (1000 ng/ml).

DNase activity assay Endogenous deoxyribonuclease (DNase) activity will be measured employing a DNase Activity Assay (Orgentec Diagnostika GmbH, Mainz, Germany). A DNA-coated microplate will be incubated with plasma samples for 60 minutes. Coated DNA will be degraded in proportion to the DNase activity of the respective sample. Optical density of residual DNA will be inversely proportional to DNase activity. All assays will be performed following the manufacturer´s instructions. All measurements will be performed in duplicate. Plates will be read on a VersaMax microplate reader (Molecular Devices, Sunnyvale, CA, USA).

Polymorphonuclear (PMN) cell culture and netosis assays PMNs (i.e. mainly neutrophils) from healthy donors will be isolated with Polymorphprep (Axis-Shield, Dundee, Scotland). Erythrocytes will be lysed using a one-step lysis buffer (NH4Cl 154mmol/L, KHCO3 10mmol/L, EDTA 0.1mmol/L). The cell suspension will then be washed twice with HBSS supplemented with 10% of fetal calf serum (FBS). Isolated PMNs will be counted and resuspended at 2x10^6 cells/ml in HBSS supplemented with 10% of FBS. Cell viability will be determined by trypan blue exclusion.

Immunofluorescence staining of NETs Fixed NETs will be stained using a mouse anti-DNA Histone H1 antibody (Millipore). After incubation, a secondary donkey anti-mouse IgG antibody coupled to Alexa Fluor 555 (Invitrogen, Life Technologies, Grand Island, NY; USA) will be added. For detection of nuclear DNA, 4',6-diamidino-2-phenylindole (DAPI, Vectashield mounting medium with DAPI; Vector Laboratories, Burlingame, CA, USA) will be used. For staining of neutrophil elastase (NE) and myeloperoxidase (MPO), rabbit anti-human NE and MPO antibodies (Abcam) are used with a secondary Alexa Fluor 488 coupled donkey anti-rabbit IgG antibody (Invitrogen). Images will be obtained with an Axio Imager 2 fluorescence microscope using AxioVision (Carl Zeiss Microscopy GmbH, Göttingen, Germany).

Statistics Normally distributed data will be expressed as mean ± standard deviation (SD), otherwise median and interquartile range (IQR) will be presented. Paired Students t-test will be applied to compare normally distributed variables, otherwise Wilcoxon signed rank test will be used. Distribution of data will be tested using the Kolmogorov-Smirnov test, the Shapiro-Wilk test and histograms (data not shown). For comparison of multiple groups, one-way analysis of variance with post-hoc Scheffé-procedure will be performed. Spearman's rank correlation (rs) will be applied to calculate correlations data. Multivariate regression models will be calculated and bootstrap correction techniques will be applied. The area under the curve (AUC) of CK-MB values will be expressed in arbitrary units and be calculated employing the trapezoidal formula (10), if at least 5 consecutive values over a period of 3 days post admission were available. Bonferroni-Holm correction will be used for multiple testing. A p-value below 0.05 will be considered significant. Statistical analyses were performed using IBM SPSS Statistics 20.0 for Windows (New York, NY, USA). Figures will be generated using GraphPad Prism 5.

ELIGIBILITY:
Inclusion Criteria:

* Medical history
* Detailed clinical examination
* Electrocardiography
* Echocardiography
* Routine blood draw (differential blood count, clotting factors including fibrinogen, liver enzymes, creatine kinase (CK), CK-MB, C-reactive protein (CRP), N-terminal pro-brain natriuretic peptide (NT-proBNP), HbA1c
* Blood draw for research experiments

Exclusion Criteria:

* Patients under 18 years; auto-immune disease, immune-modulating medication, systemic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ST elevation myocardial infarction patients, who have been hospitalized in the General Hospital of Vienna since 2006 for ST-elevation acute coronary syndrome undergoing primary percutaneous coronary intervention (pPCI) with TIMI 0-1.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of SNPs of the DNase 1 and DNase gamma genes in the STE-ACS patient population compared to healthy controls | through study completion, an average of 2 years

SECONDARY OUTCOMES:
Correlation of SNPs of the DNase 1 and gamma gene with DNase activity | through study completion, an average of 2 years
Correlation of SNPs with major adverse cardiac events | through study completion, an average of 2 years
Correlation of DNAse activity with major adverse cardiac events | through study completion, an average of 2 years
Correlation of SNPs with DNA-Histone complex levels | through study completion, an average of 2 years
Correlation of SNPs with MPO-DNA complex levels | through study completion, an average of 2 years
Correlation of SNPs with dsDNA levels | through study completion, an average of 2 years
Netosis quantification in STE-ACS patients and healthy controls | through study completion, an average of 2 years

REFERENCES:
- [Background] Nichols M, Townsend N, Scarborough P, Rayner M. Trends in age-specific coronary heart disease mortality in the European Union over three decades: 1980-2009. Eur Heart J. 2013 Oct;34(39):3017-27. doi: 10.1093/eurheartj/eht159. Epub 2013 Jun 25. PMID 23801825
- [Background] Hansson GK. Inflammation, atherosclerosis, and coronary artery disease. N Engl J Med. 2005 Apr 21;352(16):1685-95. doi: 10.1056/NEJMra043430. No abstract available. PMID 15843671
- [Background] Mangold A, Alias S, Scherz T, Hofbauer M, Jakowitsch J, Panzenbock A, Simon D, Laimer D, Bangert C, Kammerlander A, Mascherbauer J, Winter MP, Distelmaier K, Adlbrecht C, Preissner KT, Lang IM. Coronary neutrophil extracellular trap burden and deoxyribonuclease activity in ST-elevation acute coronary syndrome are predictors of ST-segment resolution and infarct size. Circ Res. 2015 Mar 27;116(7):1182-92. doi: 10.1161/CIRCRESAHA.116.304944. Epub 2014 Dec 29. PMID 25547404
- [Background] Fuchs TA, Brill A, Duerschmied D, Schatzberg D, Monestier M, Myers DD Jr, Wrobleski SK, Wakefield TW, Hartwig JH, Wagner DD. Extracellular DNA traps promote thrombosis. Proc Natl Acad Sci U S A. 2010 Sep 7;107(36):15880-5. doi: 10.1073/pnas.1005743107. Epub 2010 Aug 23. PMID 20798043
- [Background] Borissoff JI, Joosen IA, Versteylen MO, Brill A, Fuchs TA, Savchenko AS, Gallant M, Martinod K, Ten Cate H, Hofstra L, Crijns HJ, Wagner DD, Kietselaer BLJH. Elevated levels of circulating DNA and chromatin are independently associated with severe coronary atherosclerosis and a prothrombotic state. Arterioscler Thromb Vasc Biol. 2013 Aug;33(8):2032-2040. doi: 10.1161/ATVBAHA.113.301627. Epub 2013 Jul 1. PMID 23818485
- [Background] Napirei M, Ludwig S, Mezrhab J, Klockl T, Mannherz HG. Murine serum nucleases--contrasting effects of plasmin and heparin on the activities of DNase1 and DNase1-like 3 (DNase1l3). FEBS J. 2009 Feb;276(4):1059-73. doi: 10.1111/j.1742-4658.2008.06849.x. Epub 2009 Jan 16. PMID 19154352
- [Background] Ueki M, Takeshita H, Fujihara J, Iida R, Yuasa I, Kato H, Panduro A, Nakajima T, Kominato Y, Yasuda T. Caucasian-specific allele in non-synonymous single nucleotide polymorphisms of the gene encoding deoxyribonuclease I-like 3, potentially relevant to autoimmunity, produces an inactive enzyme. Clin Chim Acta. 2009 Sep;407(1-2):20-4. doi: 10.1016/j.cca.2009.06.022. Epub 2009 Jun 24. PMID 19559017
- [Background] Ueki M, Kimura-Kataoka K, Takeshita H, Fujihara J, Iida R, Sano R, Nakajima T, Kominato Y, Kawai Y, Yasuda T. Evaluation of all non-synonymous single nucleotide polymorphisms (SNPs) in the genes encoding human deoxyribonuclease I and I-like 3 as a functional SNP potentially implicated in autoimmunity. FEBS J. 2014 Jan;281(1):376-90. doi: 10.1111/febs.12608. Epub 2013 Dec 10. PMID 24206041
- [Background] Kumamoto T, Kawai Y, Arakawa K, Morikawa N, Kuribara J, Tada H, Taniguchi K, Tatami R, Miyamori I, Kominato Y, Kishi K, Yasuda T. Association of Gln222Arg polymorphism in the deoxyribonuclease I (DNase I) gene with myocardial infarction in Japanese patients. Eur Heart J. 2006 Sep;27(17):2081-7. doi: 10.1093/eurheartj/ehl177. Epub 2006 Jul 28. PMID 16877481
- [Background] Crimi G, Pica S, Raineri C, Bramucci E, De Ferrari GM, Klersy C, Ferlini M, Marinoni B, Repetto A, Romeo M, Rosti V, Massa M, Raisaro A, Leonardi S, Rubartelli P, Oltrona Visconti L, Ferrario M. Remote ischemic post-conditioning of the lower limb during primary percutaneous coronary intervention safely reduces enzymatic infarct size in anterior myocardial infarction: a randomized controlled trial. JACC Cardiovasc Interv. 2013 Oct;6(10):1055-63. doi: 10.1016/j.jcin.2013.05.011. PMID 24156966